CLINICAL TRIAL: NCT00701402
Title: Survey on Time to Lipid-lowering Drug Implementation on Dyslipidemic Patients in General Practice.
Brief Title: National Survey on Dyslipidemic Patients
Acronym: PRYSME
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CFR-DUM-2007/9
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Dyslipidemia
Keywords: time to lipid-lowering drug implementation; dyslipidemic patients
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to describe the time to lipid-lowering drug implementation in the management of dyslipidemic patients, according to the cardiovascular risk level.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dyslipemia made less than 2 years
* Treated by a lipid-lowering drug
* Agree to take part in the survey

Exclusion Criteria:

* Patient included in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First three consecutive dyslipidemic patients seen by GP
Sampling Method: Probability Sample
Enrollment: 3655 (Actual)
Dates: Start 2008-06; Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
time to lipid-lowering drug implementation (immediately, treatment within a period 0-3 month and > 3 month, according to the cardiovascular risk level, (0 risk factor, 1 risk factor, 2 risk factors, ≥ 3 risk factors, secondary prevention). | Once

CONTACTS AND LOCATIONS:
Overall Officials: Alain Castaigne, Study Director — AstraZeneca
Locations (1196):
- France (1196):
  - Research Site, Abbaretz
  - Research Site, Abbeville
  - Research Site, Ablon-sur-Seine
  - Research Site, Abrest
  - Research Site, Agde
  - Research Site, Agen
  - Research Site, Ahuy
  - Research Site, Aignay-le-Duc
  - Research Site, Aigre
  - Research Site, Aigues-Mortes
  - Research Site, Aiguillon
  - Research Site, Aix-en-Othe
  - Research Site, Aix-en-Provence
  - Research Site, Aizenay
  - Research Site, Ajaccio
  - Research Site, Alban
  - Research Site, Albens
  - Research Site, Albertville
  - Research Site, Albi
  - Research Site, Alès
  - Research Site, Alfortville
  - Research Site, Alleins
  - Research Site, Allonnes
  - Research Site, Ambillou-Château
  - Research Site, Ambleteuse
  - Research Site, Amboise
  - Research Site, Amelie LES Bains Palalda
  - Research Site, Amiens
  - Research Site, Andance
  - Research Site, Andernos-les-Bains
  - Research Site, Andrézieux-Bouthéon
  - Research Site, Anduze
  - Research Site, Angers
  - Research Site, Anglet
  - Research Site, Angoulême
  - Research Site, Aniche
  - Research Site, Annecy
  - Research Site, Annoeullin
  - Research Site, Annonay
  - Research Site, Annot
  - Research Site, Antibes
  - Research Site, Antony
  - Research Site, Anzin
  - Research Site, Arcachon
  - Research Site, Argelès-Gazost
  - Research Site, Argenteuil
  - Research Site, Arles
  - Research Site, Arras
  - Research Site, Arthez-de-Béarn
  - Research Site, Artigues-près-Bordeaux
  - Research Site, Artix
  - Research Site, Arudy
  - Research Site, Arzacq-Arraziguet
  - Research Site, Asnières-sur-Seine
  - Research Site, Aspremont
  - Research Site, Athis-Mons
  - Research Site, Aubagne
  - Research Site, Aubervilliers
  - Research Site, Aubière
  - Research Site, Auby
  - Research Site, Auch
  - Research Site, Audierne
  - Research Site, Audresselles
  - Research Site, Audun-le-Roman
  - Research Site, Aulnay-sous-Bois
  - Research Site, Aumale
  - Research Site, Auray
  - Research Site, Aureilhan
  - Research Site, Aurillac
  - Research Site, Aussonne
  - Research Site, Auterive
  - Research Site, Auvers-sur-Oise
  - Research Site, Auxerre
  - Research Site, Avignon
  - Research Site, Avion
  - Research Site, Avoine
  - Research Site, Avon
  - Research Site, Azay-le-Ferron
  - Research Site, Bachant
  - Research Site, Badonviller
  - Research Site, Bages
  - Research Site, Bagneux
  - Research Site, Bagnères-de-Luchon
  - Research Site, Bagnols-sur-Cèze
  - Research Site, Baho
  - Research Site, Bailleul
  - Research Site, Bain-de-Bretagne
  - Research Site, Bais
  - Research Site, Baisieux
  - Research Site, Balaruc-les-Bains
  - Research Site, Balma
  - Research Site, Bannalec
  - Research Site, Barr
  - Research Site, Bastia
  - Research Site, Baud
  - Research Site, Bayeux
  - Research Site, Bayonne
  - Research Site, Beaumont
  - Research Site, Beaumont-de-Lomagne
  - Research Site, Beaumont-du-Périgord
  - Research Site, Beaumont-Hague
  - Research Site, Beaumont-sur-Lèze
  - Research Site, Beaune-la-Rolande
  - Research Site, Beaurains
  - Research Site, Beauvais
  - Research Site, Beauvois-en-Cambrésis
  - Research Site, Beauzelle
  - Research Site, Belfort
  - Research Site, Bellegarde-sur-Valserine
  - Research Site, Bellême
  - Research Site, Belvès
  - Research Site, Benfeld
  - Research Site, Benquet
  - Research Site, Berck
  - Research Site, Berguette
  - Research Site, Bernay
  - Research Site, Bernin
  - Research Site, Bersée
  - Research Site, Besançon
  - Research Site, Bessan
  - Research Site, Bessines
  - Research Site, Beure
  - Research Site, Beuvrages
  - Research Site, Beynes
  - Research Site, Bezons
  - Research Site, Bègles
  - Research Site, Bélâbre
  - Research Site, Bénouville
  - Research Site, Béruges
  - Research Site, Béziers
  - Research Site, Billère
  - Research Site, Biot
  - Research Site, Biscarrosse
  - Research Site, Bischheim
  - Research Site, Blangy-sur-Bresle
  - Research Site, Blanzay
  - Research Site, Blénod-lès-Pont-à-Mousson
  - Research Site, Bobigny
  - Research Site, Boën-sur-Lignon
  - Research Site, Bohars
  - Research Site, BOIS de Nefles Saint PAUL
  - Research Site, Bois-Colombes
  - Research Site, Bois-d'Arcy
  - Research Site, Bois-en-Ardres
  - Research Site, Bompas
  - Research Site, Bondues
  - Research Site, Bonifacio
  - Research Site, Bonnelles
  - Research Site, Bonnières-sur-Seine
  - Research Site, Boos
  - Research Site, Bordeaux
  - Research Site, Bordères-sur-l'Échez
  - Research Site, Bords
  - Research Site, Bormes-les-Mimosas
  - Research Site, Bornel
  - Research Site, Bosmie-l'Aiguille
  - Research Site, Bouc-Bel-Air
  - Research Site, Boucau
  - Research Site, Bouguenais
  - Research Site, Boulogne-Billancourt
  - Research Site, Boulogne-sur-Mer
  - Research Site, Bourbourg
  - Research Site, Bourbriac
  - Research Site, Bourg
  - Research Site, Bourg-de-Péage
  - Research Site, Bourg-des-Comptes
  - Research Site, Bourg-Saint-Andéol
  - Research Site, Bourges
  - Research Site, Bousse
  - Research Site, Boutigny-sur-Essonne
  - Research Site, Braine
  - Research Site, Brantôme
  - Research Site, BRAS Panon
  - Research Site, Brest
  - Research Site, Bretenoux
  - Research Site, Breteuil
  - Research Site, Bretteville-du-Grand-Caux
  - Research Site, Bretteville-l'Orgueilleuse
  - Research Site, Breuil-le-Sec
  - Research Site, Breuillet
  - Research Site, Bréhan
  - Research Site, Brétigny-sur-Orge
  - Research Site, Brignoles
  - Research Site, Brionne
  - Research Site, Brive-la-Gaillarde
  - Research Site, Broglie
  - Research Site, Bron
  - Research Site, Brou-sur-Chantereine
  - Research Site, Brouckerque
  - Research Site, Bruay-la-Buissière
  - Research Site, Bruges
  - Research Site, Bruyères-sur-Oise
  - Research Site, Burie
  - Research Site, Burnhaupt-le-Haut
  - Research Site, Bussière-Badil
  - Research Site, Cabanac-et-Villagrains
  - Research Site, Caen
  - Research Site, Cagnes-sur-Mer
  - Research Site, Cagny
  - Research Site, Cahors
  - Research Site, Cahuzac-sur-Vère
  - Research Site, Calais
  - Research Site, Calcatoggio
  - Research Site, Caluire-et-Cuire
  - Research Site, Cambo-les-Bains
  - Research Site, Cambrai
  - Research Site, Camiers
  - Research Site, Camors
  - Research Site, Campagne-lès-Hesdin
  - Research Site, Canet
  - Research Site, Cannes
  - Research Site, Cany-Barville
  - Research Site, Capbreton
  - Research Site, Capdenac-Gare
  - Research Site, Capendu
  - Research Site, Cappelle-Brouck
  - Research Site, Carcassonne
  - Research Site, Carnoules
  - Research Site, Carquefou
  - Research Site, Casteljaloux
  - Research Site, Castelnau-Magnoac
  - Research Site, Castelnaudary
  - Research Site, Castets-en-Dorthe
  - Research Site, Castillon-en-Couserans
  - Research Site, Castres
  - Research Site, Castres-Gironde
  - Research Site, Cauchy-à-la-Tour
  - Research Site, Caudry
  - Research Site, Cauro
  - Research Site, Caussade
  - Research Site, Caux
  - Research Site, Cavaillon
  - Research Site, Caveirac
  - Research Site, Cavignac
  - Research Site, Cazes-Mondenard
  - Research Site, Ceaucé
  - Research Site, Cenon
  - Research Site, Cernay
  - Research Site, Cépet
  - Research Site, Chailland
  - Research Site, Chaingy
  - Research Site, Chaleins
  - Research Site, Chalon-sur-Saône
  - Research Site, Chambéry
  - Research Site, Champagne-sur-Seine
  - Research Site, Champagnole
  - Research Site, Champdeniers-Saint-Denis
  - Research Site, Champenoux
  - Research Site, Champigneulles
  - Research Site, Champigny-sur-Marne
  - Research Site, Champs-sur-Marne
  - Research Site, Chantepie
  - Research Site, Charenton-le-Pont
  - Research Site, Charleville-Mézières
  - Research Site, Charmont-sous-Barbuise
  - Research Site, Charnay-lès-Mâcon
  - Research Site, Chartres
  - Research Site, Chartrettes
  - Research Site, Chassieu
  - Research Site, Chatte
  - Research Site, Chaudon
  - Research Site, Chauffailles
  - Research Site, Chaulnes
  - Research Site, Chaumont
  - Research Site, Chauny
  - Research Site, Chauvigny
  - Research Site, Chavannes-sur-Suran
  - Research Site, Château-Landon
  - Research Site, Château-sur-Epte
  - Research Site, Châteauroux
  - Research Site, Châtel-Censoir
  - Research Site, Châtellerault
  - Research Site, Châtenois-les-Forges
  - Research Site, Châtres-sur-Cher
  - Research Site, Chelles
  - Research Site, Chenôve
  - Research Site, Chessy
  - Research Site, Chevilly-Larue
  - Research Site, Chigny-les-Roses
  - Research Site, Chinon
  - Research Site, Choisy-le-Roi
  - Research Site, Cholet
  - Research Site, Chusclan
  - Research Site, Cires-lès-Mello
  - Research Site, Ciré-d'Aunis
  - Research Site, Clairac
  - Research Site, Clamart
  - Research Site, Clermont-Ferrand
  - Research Site, Clichy
  - Research Site, Cluny
  - Research Site, Cognac
  - Research Site, Colmar
  - Research Site, Colombiès
  - Research Site, Combles
  - Research Site, Combourg
  - Research Site, Comines
  - Research Site, Commana
  - Research Site, Communay
  - Research Site, Comps
  - Research Site, Condat-sur-Vienne
  - Research Site, Condom
  - Research Site, Conflans STE Honorine
  - Research Site, Conliège
  - Research Site, Corbas
  - Research Site, Corbeil-Essonnes
  - Research Site, Corbeilles
  - Research Site, Corbie
  - Research Site, Cordes-sur-Ciel
  - Research Site, Cormeilles-en-Parisis
  - Research Site, Cormicy
  - Research Site, Corsept
  - Research Site, Coudekerque-Branche
  - Research Site, Couffé
  - Research Site, Couilly-Pont-aux-Dames
  - Research Site, Courbevoie
  - Research Site, Courcy
  - Research Site, Cournon-d'Auvergne
  - Research Site, Courrières
  - Research Site, Cours-la-Ville
  - Research Site, Courthézon
  - Research Site, Cousolre
  - Research Site, Crach
  - Research Site, Craponne
  - Research Site, Creil
  - Research Site, Cremeaux
  - Research Site, Creysse
  - Research Site, Crécy-la-Chapelle
  - Research Site, Crépy-en-Valois
  - Research Site, Crévic
  - Research Site, Crotenay
  - Research Site, Damazan
  - Research Site, Damparis
  - Research Site, Damprichard
  - Research Site, Daoulas
  - Research Site, Deauville
  - Research Site, Denain
  - Research Site, Digne-les-Bains
  - Research Site, Dijon
  - Research Site, Dinan
  - Research Site, Divonne-les-Bains
  - Research Site, Doazit
  - Research Site, Dol-de-Bretagne
  - Research Site, Dole
  - Research Site, Dompierre-sur-Mer
  - Research Site, Donville-les-Bains
  - Research Site, Donzenac
  - Research Site, Dormans
  - Research Site, Douarnenez
  - Research Site, Draguignan
  - Research Site, Drancy
  - Research Site, Draveil
  - Research Site, Dreux
  - Research Site, Droué
  - Research Site, Dugny-sur-Meuse
  - Research Site, Dunkirk
  - Research Site, Eaubonne
  - Research Site, Eckbolsheim
  - Research Site, Embrun
  - Research Site, Enghien-les-Bains
  - Research Site, Entre DEUX
  - Research Site, Eragny SUR OISE
  - Research Site, Escaudœuvres
  - Research Site, Eschau
  - Research Site, Esternay
  - Research Site, Estrablin
  - Research Site, Eulmont
  - Research Site, Exideuil-sur-Vienne
  - Research Site, Eybens
  - Research Site, Eygalières
  - Research Site, Eymoutiers
  - Research Site, Échenoz-la-Méline
  - Research Site, Égreville
  - Research Site, Épernay
  - Research Site, Épernon
  - Research Site, Épinal
  - Research Site, Épinay-sous-Sénart
  - Research Site, Épinay-sur-Seine
  - Research Site, Épouville
  - Research Site, Équeurdreville-Hainneville
  - Research Site, Étampes
  - Research Site, Étréchy
  - Research Site, Évenos
  - Research Site, Évin-Malmaison
  - Research Site, Évry
  - Research Site, Faremoutiers
  - Research Site, Faumont
  - Research Site, Faverolles-sur-Cher
  - Research Site, Fayl-Billot
  - Research Site, Fegersheim
  - Research Site, Figeac
  - Research Site, Firminy
  - Research Site, Fitz-James
  - Research Site, Flers-en-Escrebieux
  - Research Site, Fleurance
  - Research Site, Fleury-sur-Andelle
  - Research Site, Fonsorbes
  - Research Site, Fontaine
  - Research Site, Fontaine-lès-Luxeuil
  - Research Site, Fontainebleau
  - Research Site, Fontanil-Cornillon
  - Research Site, Fontenay-le-Comte
  - Research Site, Fontenay-sous-Bois
  - Research Site, Forbach
  - Research Site, Forges-les-Eaux
  - Research Site, Fort-Mardyck
  - Research Site, Fos-sur-Mer
  - Research Site, Fouesnant
  - Research Site, Fourmies
  - Research Site, Fourqueux
  - Research Site, Frahier-et-Chatebier
  - Research Site, Fraisans
  - Research Site, Franqueville-Saint-Pierre
  - Research Site, Fresne-Saint-Mamès
  - Research Site, Frépillon
  - Research Site, Fromentine
  - Research Site, Frontenex
  - Research Site, Fruges
  - Research Site, Gambsheim
  - Research Site, Ganges
  - Research Site, Gannat
  - Research Site, Gargenville
  - Research Site, Garges-lès-Gonesse
  - Research Site, Gelos
  - Research Site, Genas
  - Research Site, Genlis
  - Research Site, Gennes
  - Research Site, Gennevilliers
  - Research Site, Gestel
  - Research Site, Gémenos
  - Research Site, Gémozac
  - Research Site, Générac
  - Research Site, Ghisonaccia
  - Research Site, Gières
  - Research Site, Gif-sur-Yvette
  - Research Site, Gimont
  - Research Site, Ginestas
  - Research Site, Givet
  - Research Site, Givors
  - Research Site, Gometz-le-Châtel
  - Research Site, Gondrecourt-le-Château
  - Research Site, Gonesse
  - Research Site, Gorron
  - Research Site, Gourdon
  - Research Site, Goussainville
  - Research Site, Gouzon
  - Research Site, Goven
  - Research Site, Gradignan
  - Research Site, Grand-Bois
  - Research Site, Grand-Champ
  - Research Site, Grand-Charmont
  - Research Site, Grande-Synthe
  - Research Site, Grane
  - Research Site, Granville
  - Research Site, Grasse
  - Research Site, Grenoble
  - Research Site, Grignols
  - Research Site, Groslay
  - Research Site, Gruson
  - Research Site, Guenrouet
  - Research Site, Guidel
  - Research Site, Guingamp
  - Research Site, Guissény
  - Research Site, Gujan-Mestras
  - Research Site, Gurgy
  - Research Site, Guyancourt
  - Research Site, Haguenau
  - Research Site, Hallencourt
  - Research Site, Hambye
  - Research Site, Hautmont
  - Research Site, Hayange
  - Research Site, Hellemmes-Lille
  - Research Site, Hellimer
  - Research Site, Hem
  - Research Site, Hendaye
  - Research Site, Hénin-Beaumont
  - Research Site, Hombourg-Haut
  - Research Site, Hondeghem
  - Research Site, Hondschoote
  - Research Site, Houilles
  - Research Site, Hyères
  - Research Site, Hœnheim
  - Research Site, Ifs
  - Research Site, Igoville
  - Research Site, Illfurth
  - Research Site, Ingré
  - Research Site, Inzinzac-Lochrist
  - Research Site, Isbergues
  - Research Site, Isigny-le-Buat
  - Research Site, Isigny-sur-Mer
  - Research Site, Issoudun
  - Research Site, Issy-les-Moulineaux
  - Research Site, Ivry-sur-Seine
  - Research Site, Jacou
  - Research Site, Jaujac
  - Research Site, Javerlhac Chapelle Saint ROB
  - Research Site, Jenlain
  - Research Site, Jort
  - Research Site, Jouy-le-Châtel
  - Research Site, Jussey
  - Research Site, Juvigny-sous-Andaine
  - Research Site, L Etang SALE LES Bains
  - Research Site, L'Ardoise
  - Research Site, L'Escarène
  - Research Site, L'Haÿ-les-Roses
  - Research Site, L'Isle-en-Dodon
  - Research Site, L'Isle-Jourdain
  - Research Site, L'Île-Rousse
  - Research Site, L'Île-Saint-Denis
  - Research Site, La Bassée
  - Research Site, La Bastide-Clairence
  - Research Site, La Baule-Escoublac
  - Research Site, La Bazoge
  - Research Site, La Bâtie-Neuve
  - Research Site, La Bâtie-Rolland
  - Research Site, La Bernerie-en-Retz
  - Research Site, La Bouilladisse
  - Research Site, La Bouille
  - Research Site, La Brède
  - Research Site, La Buisse
  - Research Site, La Cambe
  - Research Site, La Celle-Saint-Cloud
  - Research Site, La Chapelle-Basse-Mer
  - Research Site, La Chapelle-en-Serval
  - Research Site, La Chapelle-sur-Erdre
  - Research Site, La Chèze
  - Research Site, La Ciotat
  - Research Site, La Colle-sur-Loup
  - Research Site, La Courneuve
  - Research Site, La Crau
  - Research Site, La Ferté-Frênel
  - Research Site, La Ferté-Gaucher
  - Research Site, La Fère
  - Research Site, La Fresnais
  - Research Site, La Garde
  - Research Site, La Madeleine
  - Research Site, La Mézière
  - Research Site, La Mure
  - Research Site, La Neuville-Roy
  - Research Site, La Peyrade
  - Research Site, LA Plaine DES Palmistes
  - Research Site, La Regrippière
  - Research Site, La Rivière-Saint-Sauveur
  - Research Site, La Rochelle
  - Research Site, La Rochette
  - Research Site, LA Saline LES Bains
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Source
  - Research Site, La Trimouille
  - Research Site, La Varenne-Saint-Hilaire
  - Research Site, La Verpillière
  - Research Site, La Voulte-sur-Rhône
  - Research Site, Laboutarie
  - Research Site, Lacroix-Falgarde
  - Research Site, Lagny-sur-Marne
  - Research Site, Laguépie
  - Research Site, Lambersart
  - Research Site, Lambesc
  - Research Site, Lambres
  - Research Site, Lamontjoie
  - Research Site, Lamorlaye
  - Research Site, Lampaul-Guimiliau
  - Research Site, Landéan
  - Research Site, Landébia
  - Research Site, Landévant
  - Research Site, Langlade
  - Research Site, Langoiran
  - Research Site, Langres
  - Research Site, Lansargues
  - Research Site, Lanvollon
  - Research Site, Laon
  - Research Site, Lapalud
  - Research Site, Lapeyrouse-Fossat
  - Research Site, Larche
  - Research Site, Lardy
  - Research Site, Laroquebrou
  - Research Site, Lassigny
  - Research Site, Lattes
  - Research Site, Laval
  - Research Site, Lavelanet
  - Research Site, Laveline-devant-Bruyères
  - Research Site, Laxou
  - Research Site, Le Barcarès
  - Research Site, Le Barp
  - Research Site, Le Bourg-d'Oisans
  - Research Site, Le Breuil-en-Auge
  - Research Site, Le Cannet
  - Research Site, Le Cap D'Agde
  - Research Site, Le Châtelet-en-Brie
  - Research Site, Le Cheylard
  - Research Site, Le Crès
  - Research Site, LE Guillaume
  - Research Site, Le Havre
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Langon
  - Research Site, Le Lavandou
  - Research Site, Le Mans
  - Research Site, Le Mesnil-Esnard
  - Research Site, Le Monastier-sur-Gazeille
  - Research Site, Le Nouvion-en-Thiérache
  - Research Site, Le Palais-sur-Vienne
  - Research Site, Le Pecq
  - Research Site, Le Perray-en-Yvelines
  - Research Site, Le Perreux-sur-Marne
  - Research Site, Le Pertre
  - Research Site, Le Plessis-Bouchard
  - Research Site, Le Plessis-Brion
  - Research Site, Le Plessis-Robinson
  - Research Site, Le Pont-de-Claix
  - Research Site, Le Port
  - Research Site, Le Raincy
  - Research Site, Le Relecq-Kerhuon
  - Research Site, Le Sap
  - Research Site, Le Trait
  - Research Site, Le Vaudreuil
  - Research Site, Le Verger
  - Research Site, Lecci
  - Research Site, LES Avirons
  - Research Site, Les Clayes-sous-Bois
  - Research Site, Les Epesses
  - Research Site, Les Gonds
  - Research Site, Les Lilas
  - Research Site, Les Loges
  - Research Site, Les Lucs-sur-Boulogne
  - Research Site, Les Mureaux
  - Research Site, Les Paroches
  - Research Site, Les Pennes-Mirabeau
  - Research Site, Les Sables-d'Olonne
  - Research Site, Lesconil
  - Research Site, Lesquin
  - Research Site, Levallois-Perret
  - Research Site, Lège-Cap-Ferret
  - Research Site, Léry
  - Research Site, Liévin
  - Research Site, Ligny-le-Ribault
  - Research Site, Lille
  - Research Site, Lillebonne
  - Research Site, Limoges
  - Research Site, Limoux
  - Research Site, Lixing-lès-Saint-Avold
  - Research Site, Lognes
  - Research Site, Lombron
  - Research Site, Lomme
  - Research Site, Longeville-lès-Saint-Avold
  - Research Site, Longpont-sur-Orge
  - Research Site, Longueau
  - Research Site, Loos
  - Research Site, Loperhet
  - Research Site, Lormont
  - Research Site, Lorrez-le-Bocage-Préaux
  - Research Site, Louverné
  - Research Site, Louvigné-du-Désert
  - Research Site, Louvroil
  - Research Site, Luçay-le-Mâle
  - Research Site, Luçon
  - Research Site, Lunel
  - Research Site, Lunery
  - Research Site, Lunéville
  - Research Site, Lure
  - Research Site, Lusignan
  - Research Site, Luz-Saint-Sauveur
  - Research Site, Luzarches
  - Research Site, Lyon
  - Research Site, Machecoul
  - Research Site, Magagnosc
  - Research Site, Magny-en-Vexin
  - Research Site, Maisons-Alfort
  - Research Site, Maizières-lès-Metz
  - Research Site, Malakoff
  - Research Site, Malesherbes
  - Research Site, Malestroit
  - Research Site, Malicorne-sur-Sarthe
  - Research Site, Mandelieu-la-Napoule
  - Research Site, Mandeure
  - Research Site, Manosque
  - Research Site, Mansac
  - Research Site, Mantes-la-Jolie
  - Research Site, Mantes-la-Ville
  - Research Site, Marcigny
  - Research Site, Marcoussis
  - Research Site, Marcq-en-Barœul
  - Research Site, Mareuil
  - Research Site, Marignane
  - Research Site, Marles-les-Mines
  - Research Site, Marly
  - Research Site, Marquette-lez-Lille
  - Research Site, Marquillies
  - Research Site, Marquise
  - Research Site, Marseille
  - Research Site, Martigny-les-Bains
  - Research Site, Martigues
  - Research Site, Masnières
  - Research Site, Mauguio
  - Research Site, Maurecourt
  - Research Site, Maurepas
  - Research Site, Mayenne
  - Research Site, Mayet
  - Research Site, Mâcon
  - Research Site, Meaux
  - Research Site, Megève
  - Research Site, Meistratzheim
  - Research Site, Melun
  - Research Site, Menthon-Saint-Bernard
  - Research Site, Menton
  - Research Site, Merlevenez
  - Research Site, Messia-sur-Sorne
  - Research Site, Metz
  - Research Site, Meursault
  - Research Site, Meylan
  - Research Site, Meyssac
  - Research Site, Méjannes-lès-Alès
  - Research Site, Méounes-lès-Montrieux
  - Research Site, Mérignac
  - Research Site, Méru
  - Research Site, Méry-sur-Seine
  - Research Site, Mézières-en-Brenne
  - Research Site, Migennes
  - Research Site, Millas
  - Research Site, Mimet
  - Research Site, Mimizan
  - Research Site, Miramas
  - Research Site, Mirambeau
  - Research Site, Miribel
  - Research Site, Mittelhausen
  - Research Site, Molinghem
  - Research Site, Molsheim
  - Research Site, Moncontour de Bretagne
  - Research Site, Mondragon
  - Research Site, Monistrol-sur-Loire
  - Research Site, Mont-Saint-Martin
  - Research Site, Mont-sous-Vaudrey
  - Research Site, Montady
  - Research Site, Montargis
  - Research Site, Montauban
  - Research Site, Montauban-de-Bretagne
  - Research Site, Montbeton
  - Research Site, Montbrison
  - Research Site, Montceau-les-Mines
  - Research Site, Monterblanc
  - Research Site, Montereau-Fault-Yonne
  - Research Site, Monteux
  - Research Site, Montfaucon-d'Argonne
  - Research Site, Montfermeil
  - Research Site, Montfort-sur-Meu
  - Research Site, Montgeron
  - Research Site, Montigny-lès-Cormeilles
  - Research Site, Montlignon
  - Research Site, Montmagny
  - Research Site, Montmorillon
  - Research Site, Montoire-sur-le-Loir
  - Research Site, Montpellier
  - Research Site, Montpon-Ménestérol
  - Research Site, Montreuil
  - Research Site, Montreuil-Bellay
  - Research Site, Montréjeau
  - Research Site, Montrouge
  - Research Site, Montry
  - Research Site, Moosch
  - Research Site, Mornas
  - Research Site, Mortagne-du-Nord
  - Research Site, Mortain
  - Research Site, Morteau
  - Research Site, Moufia
  - Research Site, Mougins
  - Research Site, Moulins
  - Research Site, Moussy-le-Neuf
  - Research Site, Mouvaux
  - Research Site, Moûtiers
  - Research Site, Moyaux
  - Research Site, Mozac
  - Research Site, Mulhouse
  - Research Site, Muntzenheim
  - Research Site, Muret
  - Research Site, Murviel-lès-Béziers
  - Research Site, Mussig
  - Research Site, Nancray
  - Research Site, Nancy
  - Research Site, Nantes
  - Research Site, Narbonne
  - Research Site, Navarrenx
  - Research Site, Neufchâtel-sur-Aisne
  - Research Site, Neuilly-l'Évêque
  - Research Site, Neuilly-sur-Marne
  - Research Site, Neuvic
  - Research Site, Neuville-lès-Dieppe
  - Research Site, Neuville-sur-Sarthe
  - Research Site, Nevers
  - Research Site, Nexon
  - Research Site, Nérac
  - Research Site, Nice
  - Research Site, Nieul-sur-Mer
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Nods
  - Research Site, Nogent-le-Rotrou
  - Research Site, Nogent-sur-Aube
  - Research Site, Noisiel
  - Research Site, Noisy-le-Grand
  - Research Site, Nommay
  - Research Site, Notre-Dame-d'Oé
  - Research Site, Notre-Dame-de-Gravenchon
  - Research Site, Notre-Dame-du-Touchet
  - Research Site, Nouzonville
  - Research Site, Novalaise
  - Research Site, Novéant-sur-Moselle
  - Research Site, Noyal-Châtillon-sur-Seiche
  - Research Site, Noyant
  - Research Site, Noyant-la-Gravoyère
  - Research Site, Noyon
  - Research Site, Octeville
  - Research Site, Oissel-sur-Seine
  - Research Site, Ollioules
  - Research Site, Oradour-sur-Vayres
  - Research Site, Orange
  - Research Site, Orchies
  - Research Site, Orléans
  - Research Site, Orvault
  - Research Site, Ostwald
  - Research Site, Oullins
  - Research Site, Outreau
  - Research Site, Oyonnax
  - Research Site, Ozoir-la-Ferrière
  - Research Site, Paillencourt
  - Research Site, Palaiseau
  - Research Site, Palau-del-Vidre
  - Research Site, Panissières
  - Research Site, Pantin
  - Research Site, Parçay-les-Pins
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Peaugres
  - Research Site, Pecquencourt
  - Research Site, Perpignan
  - Research Site, Perrigny
  - Research Site, Perros-Guirec
  - Research Site, Pertuis
  - Research Site, Pessac
  - Research Site, Petit-Couronne
  - Research Site, Petit-Mars
  - Research Site, Petite ILE
  - Research Site, Peujard
  - Research Site, Peyruis
  - Research Site, Pépieux
  - Research Site, Périgueux
  - Research Site, Pfastatt
  - Research Site, Pfulgriesheim
  - Research Site, Pierre-Bénite
  - Research Site, Pierre-Buffière
  - Research Site, Pierrefonds
  - Research Site, Pisany
  - Research Site, Plaisance
  - Research Site, Pleaux
  - Research Site, Pleumeur-Bodou
  - Research Site, Pleyber-Christ
  - Research Site, Ploubezre
  - Research Site, Plouër-sur-Rance
  - Research Site, Ploufragan
  - Research Site, Plouvien
  - Research Site, Poillé-sur-Vègre
  - Research Site, Poitiers
  - Research Site, Poligny
  - Research Site, Poncin
  - Research Site, Pont du Fossé
  - Research Site, PONT STE Maxence
  - Research Site, Pont-de-Buis-lès-Quimerch
  - Research Site, Pont-l'Évêque
  - Research Site, Pontacq
  - Research Site, Pontailler-sur-Saône
  - Research Site, Pontault-Combault
  - Research Site, Pontcharra-sur-Turdine
  - Research Site, Ponte Leccia
  - Research Site, Pontoise
  - Research Site, Pornic
  - Research Site, Port-sur-Saône
  - Research Site, Potigny
  - Research Site, Pouilly-sur-Loire
  - Research Site, Pourrières
  - Research Site, Poussan
  - Research Site, Pradines
  - Research Site, Prat
  - Research Site, Prémery
  - Research Site, Puttelange-aux-Lacs
  - Research Site, Puylaurens
  - Research Site, Quimper
  - Research Site, Quint-Fonsegrives
  - Research Site, Ramonville-Saint-Agne
  - Research Site, Ravine DES Cabris
  - Research Site, Râches
  - Research Site, Reims
  - Research Site, Reiningue
  - Research Site, Revel
  - Research Site, Réalville
  - Research Site, Rémilly
  - Research Site, Ribeauvillé
  - Research Site, Rieumes
  - Research Site, Rion-des-Landes
  - Research Site, Riorges
  - Research Site, Ris-Orangis
  - Research Site, Rixheim
  - Research Site, Roanne
  - Research Site, Robert-Espagne
  - Research Site, Robion
  - Research Site, Rochefort-du-Gard
  - Research Site, Rochefort-en-Terre
  - Research Site, Rognes
  - Research Site, Romainville
  - Research Site, Romorantin-Lanthenay
  - Research Site, Ronchin
  - Research Site, Roquebrune-Cap-Martin
  - Research Site, Rosendaël
  - Research Site, Rosny-sous-Bois
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Rouillac
  - Research Site, Royan
  - Research Site, Roye
  - Research Site, Rozérieulles
  - Research Site, Rueil-Malmaison
  - Research Site, Rungis
  - Research Site, Sablé-sur-Sarthe
  - Research Site, Saillans
  - Research Site, Sainpuits
  - Research Site, Saint Denis Chaudron
  - Research Site, Saint Gilles LES Hauts
  - Research Site, Saint Maximin LA STE Baume
  - Research Site, Saint-Agrève
  - Research Site, Saint-Aignan
  - Research Site, Saint-Amand-sur-Sèvre
  - Research Site, Saint-Andiol
  - Research Site, Saint-André-d'Apchon
  - Research Site, Saint-André-de-Cubzac
  - Research Site, Saint-André-les-Vergers
  - Research Site, Saint-André-lez-Lille
  - Research Site, Saint-Augustin
  - Research Site, Saint-Benoît
  - Research Site, Saint-Briac-sur-Mer
  - Research Site, Saint-Brice-sous-Forêt
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Chamond
  - Research Site, Saint-Chéron
  - Research Site, Saint-Cloud
  - Research Site, Saint-Cyr-sur-Loire
  - Research Site, Saint-Denis
  - Research Site, Saint-Dizier
  - Research Site, Saint-Etienne
  - Research Site, Saint-Émilion
  - Research Site, Saint-Étienne-de-Montluc
  - Research Site, Saint-Étienne-du-Rouvray
  - Research Site, Saint-Étienne-lès-Remiremont
  - Research Site, Saint-Féliu-d'Avall
  - Research Site, Saint-Florent-des-Bois
  - Research Site, Saint-Geniès-Bellevue
  - Research Site, Saint-Georges-de-Reneins
  - Research Site, Saint-Georges-sur-Baulche
  - Research Site, Saint-Germain-au-Mont-d'Or
  - Research Site, Saint-Germain-de-la-Coudre
  - Research Site, Saint-Gervais-la-Forêt
  - Research Site, Saint-Girons
  - Research Site, Saint-Glen
  - Research Site, Saint-Gratien
  - Research Site, Saint-Herblain
  - Research Site, Saint-Hilaire-de-Riez
  - Research Site, Saint-Hilaire-lez-Cambrai
  - Research Site, Saint-Jean-de-la-Ruelle
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Saint-Jorioz
  - Research Site, Saint-Joseph
  - Research Site, Saint-Julien-en-Genevois
  - Research Site, Saint-Julien-le-Faucon
  - Research Site, Saint-Julien-les-Villas
  - Research Site, Saint-Just-Saint-Rambert
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Saint-Leu
  - Research Site, Saint-Leu-d'Esserent
  - Research Site, Saint-Leu-la-Forêt
  - Research Site, Saint-Léger-des-Bois
  - Research Site, Saint-Léger-en-Yvelines
  - Research Site, Saint-Louis
  - Research Site, Saint-Lys
  - Research Site, Saint-Marcel
  - Research Site, Saint-Martin-Bellevue
  - Research Site, Saint-Martin-Boulogne
  - Research Site, Saint-Martin-d'Oney
  - Research Site, Saint-Martin-d'Uriage
  - Research Site, Saint-Martin-de-Crau
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Martin-des-Noyers
  - Research Site, Saint-Martin-en-Haut
  - Research Site, Saint-Martin-le-Vinoux
  - Research Site, Saint-Martin-sur-le-Pré
  - Research Site, Saint-Maur-des-Fossés
  - Research Site, Saint-Maurice-sur-Aveyron
  - Research Site, Saint-Max
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Nectaire
  - Research Site, Saint-Omer
  - Research Site, Saint-Ouen
  - Research Site, Saint-Pardoux
  - Research Site, Saint-Pathus
  - Research Site, Saint-Paul-lès-Dax
  - Research Site, Saint-Pierre-d'Albigny
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Pol-de-Léon
  - Research Site, Saint-Prest
  - Research Site, Saint-Quentin
  - Research Site, Saint-Rambert-en-Bugey
  - Research Site, Saint-Raphaël
  - Research Site, Saint-Rémy-de-Provence
  - Research Site, Saint-Saulve
  - Research Site, Saint-Sauveur-en-Puisaye
  - Research Site, Saint-Sébastien-sur-Loire
  - Research Site, Saint-Sylvain
  - Research Site, Saint-Symphorien-sur-Coise
  - Research Site, Saint-Thibéry
  - Research Site, Saint-Vincent-de-Tyrosse
  - Research Site, Saint-Yorre
  - Research Site, Sainte-Geneviève-des-Bois
  - Research Site, Salmiech
  - Research Site, Sarcelles
  - Research Site, Sarlat-la-Canéda
  - Research Site, Sarras
  - Research Site, Sarreguemines
  - Research Site, Sarry
  - Research Site, Sartrouville
  - Research Site, Saulon-la-Chapelle
  - Research Site, Sausset-les-Pins
  - Research Site, Sauvagnon
  - Research Site, Sauzé-Vaussais
  - Research Site, Saverne
  - Research Site, Savigneux
  - Research Site, Savigné-l'Évêque
  - Research Site, Savigny-sur-Orge
  - Research Site, Scey-sur-Saône-et-Saint-Albin
  - Research Site, Schiltigheim
  - Research Site, Seclin
  - Research Site, Selles-sur-Cher
  - Research Site, Semur-en-Auxois
  - Research Site, Sens
  - Research Site, Sercœur
  - Research Site, Serres
  - Research Site, Servins
  - Research Site, Sète
  - Research Site, Sées
  - Research Site, Sigean
  - Research Site, Sillery
  - Research Site, Sillé-le-Guillaume
  - Research Site, Sochaux
  - Research Site, Soissons
  - Research Site, Somain
  - Research Site, Sorbiers
  - Research Site, Sorcy-Saint-Martin
  - Research Site, Sotteville-lès-Rouen
  - Research Site, Soucieu-en-Jarrest
  - Research Site, Soueich
  - Research Site, Souillac
  - Research Site, Soulac-sur-Mer
  - Research Site, Soultz-sous-Forêts
  - Research Site, Souppes-sur-Loing
  - Research Site, Soyons
  - Research Site, Spéracèdes
  - Research Site, St Chamas
  - Research Site, St-Malo
  - Research Site, STE Adresse
  - Research Site, STE Clotilde
  - Research Site, STE Eulalie
  - Research Site, STE Gemmes SUR Loire
  - Research Site, STE Marie de RE
  - Research Site, STE Marie
  - Research Site, STE Sigolene
  - Research Site, STE Suzanne
  - Research Site, Strasbourg
  - Research Site, Surgères
  - Research Site, Taillades
  - Research Site, Talence
  - Research Site, Tantonville
  - Research Site, Tence
  - Research Site, Ternay
  - Research Site, Terre Sainte
  - Research Site, Terville
  - Research Site, Theix
  - Research Site, Thénezay
  - Research Site, Thiaucourt-Regniéville
  - Research Site, Thiers
  - Research Site, Thionville
  - Research Site, Thiviers
  - Research Site, Thoirette
  - Research Site, Thoré-la-Rochette
  - Research Site, Thorigny-sur-Oreuse
  - Research Site, Thouaré-sur-Loire
  - Research Site, Thouars
  - Research Site, Tilloy-lès-Mofflaines
  - Research Site, Tinqueux
  - Research Site, Tonnerre
  - Research Site, Tosse
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tourlaville
  - Research Site, Tournon-sur-Rhône
  - Research Site, Tourrettes-sur-Loup
  - Research Site, Tours
  - Research Site, Travo
  - Research Site, Treillières
  - Research Site, Tremblay
  - Research Site, Trégourez
  - Research Site, Troisfontaines
  - Research Site, Troyes
  - Research Site, Tulle
  - Research Site, Uchaud
  - Research Site, Uckange
  - Research Site, Uriage-les-Bains
  - Research Site, Urzy
  - Research Site, Usson-en-Forez
  - Research Site, Vailhauquès
  - Research Site, Vairé
  - Research Site, Vaison-la-Romaine
  - Research Site, Val-de-Vesle
  - Research Site, Valdahon
  - Research Site, Valence
  - Research Site, Valence-d'Albigeois
  - Research Site, Valergues
  - Research Site, Vallabrègues
  - Research Site, Vallauris
  - Research Site, Valleiry
  - Research Site, Valleraugue
  - Research Site, Valognes
  - Research Site, Valras-Plage
  - Research Site, Valréas
  - Research Site, Vanault-les-Dames
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vannes
  - Research Site, Varangéville
  - Research Site, Varennes
  - Research Site, Varennes-Vauzelles
  - Research Site, Vasles
  - Research Site, Vaucresson
  - Research Site, Vauhallan
  - Research Site, Vaulx-en-Velin
  - Research Site, Vaux-le-Pénil
  - Research Site, Vedène
  - Research Site, Verberie
  - Research Site, Verfeil
  - Research Site, Vern-sur-Seiche
  - Research Site, Verneuil-sur-Seine
  - Research Site, Vers-Pont-du-Gard
  - Research Site, Versailles
  - Research Site, Vertou
  - Research Site, Verzy
  - Research Site, Vesoul
  - Research Site, Vézelise
  - Research Site, Vic-la-Gardiole
  - Research Site, Vichy
  - Research Site, Vienne
  - Research Site, Vignacourt
  - Research Site, Vigneux-sur-Seine
  - Research Site, Villabé
  - Research Site, Villars-les-Dombes
  - Research Site, Ville-la-Grand
  - Research Site, Villebon-sur-Yvette
  - Research Site, Villefranche-de-Lonchat
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villemomble
  - Research Site, Villenave-d'Ornon
  - Research Site, Villeneuve-la-Comtesse
  - Research Site, Villeneuve-Saint-Georges
  - Research Site, Villepreux
  - Research Site, Villerest
  - Research Site, Villers-Bretonneux
  - Research Site, Villers-Cotterêts
  - Research Site, Villers-lès-Nancy
  - Research Site, Villers-Outréaux
  - Research Site, Villers-Saint-Paul
  - Research Site, Villette-d'Anthon
  - Research Site, Villeurbanne
  - Research Site, Villeveyrac
  - Research Site, Villey-Saint-Étienne
  - Research Site, Villiers-sur-Marne
  - Research Site, Villiers-sur-Orge
  - Research Site, Vincennes
  - Research Site, Vinça
  - Research Site, Vire
  - Research Site, Viriville
  - Research Site, Vitré
  - Research Site, Vitrolles
  - Research Site, Vitry-sur-Seine
  - Research Site, Vittefleur
  - Research Site, Viviers
  - Research Site, Voiron
  - Research Site, Vouillé
  - Research Site, Voujeaucourt
  - Research Site, Wambrechies
  - Research Site, Wasselonne
  - Research Site, Wattrelos
  - Research Site, Waziers
  - Research Site, Wingles
  - Research Site, Wissant
  - Research Site, Yquelon